CLINICAL TRIAL: NCT06324331
Title: The Impact of Decidual al Sparing During Uterine Closure on Post Cesarean Niche Formation
Brief Title: Effect of Decidual Sparing in cs Niche Formation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna Allah Abd Elaziaz Ahmed, Resident, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: Decidual sparing & CS niche
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section Complications; Cesarean Section Niche
Keywords: Decidual sparing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non decidual sparing (Experimental): uterine incision repair including suturing of the endometrium
  Interventions: Procedure: Non decidual sparing
- Decidual sparing (Experimental): uterine incision repair without including the endometrium.
  Interventions: Procedure: Decidual sparing

INTERVENTIONS:
Procedure: Decidual sparing — Endometrial free uterine closure technique
  Arms: Decidual sparing
Procedure: Non decidual sparing — Routine uterine closure technique including endometrium
  Arms: Non decidual sparing

SUMMARY:
Assessing the impact of endometrial sparing at double-layer uterine closure as a specific surgical technique in CS to reduce the rate of post-cessarian delivery niche develoment

DETAILED DESCRIPTION:
A Cesarean scar defect (CSD) or niche, also termed isthmocele, has been the subject of intensive research over the past 20 years, which resulted in over 3000 publications worldwide. At the beginning of the twentieth century, a cesarean scar described as furrow was noted in hysterectomized uteri of women after a Cesarean delivery (CD). In 2001, Monteagudo et al. described a specific intrauterine defect or niche, using saline infusion sonohysterography (SIS), as a triangular hypoechoic/ anechoic fluid-filled space present in uteri of 40 women with postmenopausal bleeding who had a previous cesarean delivery, reflecting a discontinuity of the myometrium at the site of the uterine incision scar, most likely the result of incomplete healing.The degree of defect, referring to the size of the niche and the thinness of the residual myometrial thickness (RMT) by ultrasound, is often associated with a higher complication rate. The presence of a niche is associated with other dangerous obstetrical complications, such as Cesarean scar pregnancies (CSP), placenta accreta spectrum (PAS), as well as numerous gynecological problems, including intermenstrual spotting, dysmenorrhea, pelvic pain, subfertility, and suboptimal IVF implantation rate.3As the absolute number of CDs increased, their associated complications presented significant challenges for patients, providers, and researchers. Several hypotheses have been advanced to explain niche formation, including oxygen deprivation, poor tissue healing, surgical techniques, and maternal factors.A recent publication described the origin of a post-CD niche following uterine closure. The authors outlined the uterine defect immediately by SIS and, using histopathological studies, demonstrated the presence of the decidua lining the defect, extending, and penetrating the surface of the incision. The inclusion of the endometrium into the uterine closure and lack of myometrial approximation were video recorded.Although these findings have implications for layer-to-layer approximation, the clinical relevance of niche development remains unclear, as its association with intrinsic surgical techniques remains poorly investigated. Possible reasons: Most studies include heterogeneous groups of patients, surgeons, and uterine closure techniques offering no uniform understanding of niche development and size. Reading the history of uterine closure techniques, in 1882, Max Sänger cautioned to avoid the decidua into the uterine closure of the classical cesarean operation, which has become the present-day classical CS8 . The practice of avoiding including the decidua into the uterine wall closure was taught and practiced until the 1970s, gradually losing popularity as newer closure techniques were described.10-12 These more recent developments made no reference to how to handle the endometrium during incision closure. The impact of the endometrium on scar strength and integrity has been studied in animal and human models.A recent retrospective study of 4496 consecutive deliveries was conducted and concluded that there was no abnormal placentation in subsequent pregnancies of 737 women who underwent a CD during the 30-year period when a specific technique termed endometrium-free uterine closure technique (EFCT) was employed16 . This study compares the incidence and size of uterine niches after routine closure technique of the CD incision versus the EFCT using TVUS in their non-pregnant state among women with one prior CD.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy of gestational age ≥ 32wks

Exclusion Criteria:

* previous uterine scar

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Impact of decidual sparing on niche formation | 3-6 months post CS
  Assessing incidence of niche formation in EFCT vs routine uterine closure of CS by TVUS

SECONDARY OUTCOMES:
Impact of uterine closure technique on post CS niche criteria | 3-6 months post CS
  the size of the niche defect measured by depth, width, length, and RMT above its apex